CLINICAL TRIAL: NCT02564029
Title: A Double Blind, Randomized, Cross- Over Study Examining Efficacy Of Pf-06372865 In A Photosensitivity Epilepsy Study Using Lorazepam As A Positive Control
Brief Title: PF-06372865 in Subjects With Photosensitive Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B7431005
Record Dates: First submitted 2015-09-10; First posted 2015-09-30 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: Reflex Epilepsy, Photosensitive
MeSH Terms: conditions — Epilepsy, Reflex | interventions — PF-06372865; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-06372865 dose level 1 (Experimental): 17.5 milligram (mg) single dose
  Interventions: Drug: PF-06372865
- PF-06372865 dose level 2 (Experimental): 52.5 mg single dose
  Interventions: Drug: PF-06372865
- Placebo (Placebo Comparator): Single dose
  Interventions: Drug: Placebo
- Lorazepam (Active Comparator): 2mg single dose
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: PF-06372865 — Single dose
  Arms: PF-06372865 dose level 1; PF-06372865 dose level 2
Drug: Placebo — Placebo for PF-06372865 and placebo for lorazepam
  Arms: Placebo
Drug: Lorazepam — 2 mg single oral dose
  Arms: Lorazepam

SUMMARY:
PF-06372865 in subjects with photosensitive epilepsy

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis and history of photoparoxysmal response on electroencephalogram (EEG) with or without a diagnosis of epilepsy for which subjects are taking up to 0 - 2 concomitant antiepileptic drugs.
* Subjects currently taking antiepileptic drug(s) to be on a stable dose for 4 weeks prior to Screening Visit.
* A minimum average standardized photosensitive range (SPR) across all screening timepoints of 4 in the most sensitive eye condition and a non-zero average in at least one other eye condition.

Exclusion Criteria:

* Subjects with a history of status epilepticus.
* Subjects who have experienced a generalized tonic-clonic convulsion in the past 6 months, at the time of the initial screening visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Consultants in Epilepsy & Neurology, PLLC, Boise, Idaho
  - Johns Hopkins University Department of Neurology, Baltimore, Maryland
  - Barnes Jewish Hospital, St Louis, Missouri
  - Center for Advanced Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - New York University Comprehensive Epilepsy Center, New York, New York
  - Clinical and Translational Research Center, Philadelphia, Pennsylvania
  - Hospital of the Univ of PA Pharmacy Service, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Comprehensive Epilepsy Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital EEG lab, Philadelphia, Pennsylvania
  - Thomas Jefferson University Investigational Drug Service, Philadelphia, Pennsylvania
  - General Clinical Research Center (GCRC), Nashville, Tennessee
  - Vanderbilt University Epilepsy Clinic, Nashville, Tennessee
  - Vanderbilt University Hospital Pharmacy, Nashville, Tennessee
  - VU Department of Neurology, Nashville, Tennessee

REFERENCES:
- [Derived] Gurrell R, Gorman D, Whitlock M, Ogden A, Reynolds DS, DiVentura B, Abou-Khalil B, Gelfand M, Pollard J, Hogan RE, Krauss G, Sperling M, Vazquez B, Wechsler RT, Friedman D, Butt RP, French J. Photosensitive epilepsy: Robust clinical efficacy of a selective GABA potentiator. Neurology. 2019 Apr 9;92(15):e1786-e1795. doi: 10.1212/WNL.0000000000007271. Epub 2019 Mar 15. PMID 30877186
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7431005&StudyName=A%20Double%20Blind%2C%20Randomized%2C%20Cross-%20Over%20Study%20Examining%20Efficacy%20Of%20Pf-06372865%20In%20A%20Photosensitivity%20Epilepsy%20Study%20Using%20Lorazepam%20As%20A%20Positive%20Control

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Subjects were randomly allocated to one of 4 different treatment sequences that each included the 4 treatment groups: Placebo, PF-06372865 17.5 mg, PF-06372865 52.5 mg and Lorazepam 2 mg.
Period: Overall Study
Arm/Group | All Study Participants
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: all participants randomized and who had received at least 1 dose of randomized treatment and had at least 1 primary efficacy measurement in at least 1 study treatment period.
Groups:
- All Participants: A total of 7 participants were enrolled and assigned to study treatment.
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Standardized Photosensitivity Range (SPR) in the Subject's Most Sensitive Eye Condition
Description: The SPR was defined as the number of frequency steps between and including the lower and upper bound at which a generalized electroencephalogram (EEG) epileptiform activity had occurred, whereby subjects were exposed to 14 different frequencies ranging from 2 to 60 flashes per second. The SPR is then an integer score that ranges from 0 to 14 with lower scores representing better outcomes. The primary outcome measure was based on the average Least Squares Mean (LSmean) effect over the first 6 hours postdose.
Time Frame: Pre-dose, 1, 2, 4 and 6 hours post-dose
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- PF-06372865 17.5 mg: One (1) lorazepam placebo tablet and seven (7) PF-06372865 2.5 mg tablets.
- PF-06372865 52.5 mg: One (1) lorazepam placebo tablet and seven (7) PF-06372865 7.5 mg tablets.
- Lorazepam 2 mg: One (1) lorazepam 2 mg tablet and seven (7) PF-06372865 placebo tablets.
- Placebo: One (1) lorazepam placebo tablet and seven (7) PF-06372865 placebo tablets.
Arm/Group | PF-06372865 17.5 mg | PF-06372865 52.5 mg | Lorazepam 2 mg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 7
Units on a scale | 0.57 (0.98) | 1.38 (0.96) | 1.58 (0.97) | 6.80 (0.96)
Statistical Analysis 1: Comparison: PF-06372865 17.5 mg vs Placebo; A mixed effects model was applied with fixed effects for period, time, treatment, and the interaction between treatment and time. Baseline was included as 2 separate covariates. The interaction between each baseline covariate and time were included as fixed effects. Participant was fitted as a random effect and time was fitted as a repeated effect within each participant × period. An unstructured correlation matrix was used. The effect reported is an average across all post-dose measurements; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -6.23, 90% CI 2-sided [-8.60 to -3.86], Standard Error of Mean 1.37
Statistical Analysis 2: Comparison: PF-06372865 52.5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -5.42, 90% CI 2-sided [-7.78 to -3.06], Standard Error of Mean 1.36
Statistical Analysis 3: Comparison: Lorazepam 2 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -5.22, 90% CI 2-sided [-7.60 to -2.84], Standard Error of Mean 1.37
Statistical Analysis 4: Comparison: PF-06372865 17.5 mg vs PF-06372865 52.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = 0.81, 90% CI 2-sided [-1.58 to 3.20], Standard Error of Mean 1.38
Statistical Analysis 5: Comparison: PF-06372865 17.5 mg vs Lorazepam 2 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mixed Model Repreated Measure Analysis; Mean Difference (Final Values) = -1.01, 90% CI 2-sided [-3.43 to 1.41], Standard Error of Mean 1.4
Statistical Analysis 6: Comparison: PF-06372865 52.5 mg vs Lorazepam 2 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -0.2, 90% CI 2-sided [-2.56 to 2.16], Standard Error of Mean 1.36

2. Secondary Outcome: The SPR in the Eye Closure, Eyes Closed, and Eyes Open Condition
Description: The SPR was defined as the number of frequency steps between and including the lower and upper bound at which a generalized electroencephalogram (EEG) epileptiform activity had occurred, whereby subjects were exposed to 14 different frequencies ranging from 2 to 60 flashes per second. The SPR is then an integer score that ranges from 0 to 14 with lower scores representing better outcomes. The outcome measure was based on the average Least Squares Mean (LSmean) effect over the first 6 hours postdose.
Time Frame: Pre-dose, 1, 2, 4 and 6 hours post-dose
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-06372865 17.5 mg | PF-06372865 52.5 mg | Lorazepam 2 mg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 7
Units on a scale
  Eye Closure | 0.57 (0.98) | 1.38 (0.96) | 1.58 (0.97) | 6.80 (0.96)
  Eyes Closed: number analyzed (Participants) | 7 | 7 | 7 | 6
  Eyes Closed | 0.33 (0.57) | 0.40 (0.57) | 1.09 (0.57) | 6.84 (0.64)
  Eyes Open: number analyzed (Participants) | 7 | 7 | 7 | 6
  Eyes Open | 0.04 (0.46) | 0.09 (0.46) | 0.08 (0.46) | 4.46 (0.51)
Statistical Analysis 1: Comparison: PF-06372865 17.5 mg vs Placebo; In eye closure condition. The same mixed model repeated measures analysis as applied to the primary outcome measure was used; Test type: Other; Mixed Model Repeated Measure Analysis; Mean Difference (Final Values) = -6.23, 90% CI 2-sided [-8.60 to -3.86], Standard Error of Mean 1.37
Statistical Analysis 2: Comparison: PF-06372865 52.5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -5.42, 90% CI 2-sided [-7.78 to -3.06], Standard Error of Mean 1.36
Statistical Analysis 3: Comparison: Lorazepam 2 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -5.22, 90% CI 2-sided [-7.60 to -2.84], Standard Error of Mean 1.37
Statistical Analysis 4: Comparison: PF-06372865 17.5 mg vs PF-06372865 52.5 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = 0.81, 90% CI 2-sided [-1.58 to 3.20], Standard Error of Mean 1.38
Statistical Analysis 5: Comparison: PF-06372865 17.5 mg vs Lorazepam 2 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -1.01, 90% CI 2-sided [-3.43 to 1.41], Standard Error of Mean 1.4
Statistical Analysis 6: Comparison: PF-06372865 52.5 mg vs Lorazepam 2 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -0.2, 90% CI 2-sided [-2.56 to 2.16], Standard Error of Mean 1.36
Statistical Analysis 7: Comparison: PF-06372865 17.5 mg vs Placebo; In eyes closed condition. The same mixed model repeated measures analysis as applied to the primary outcome measure was used; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -6.51, 90% CI 2-sided [-8.01 to -5.01], Standard Error of Mean 0.79
Statistical Analysis 8: Comparison: PF-06372865 52.5 mg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -6.44, 90% CI 2-sided [-7.93 to -4.95], Standard Error of Mean 0.78
Statistical Analysis 9: Comparison: Lorazepam 2 mg vs Placebo; [analysis description as in outcome 2, analysis 7]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -5.74, 90% CI 2-sided [-7.20 to -4.28], Standard Error of Mean 0.76
Statistical Analysis 10: Comparison: PF-06372865 17.5 mg vs PF-06372865 52.5 mg; [analysis description as in outcome 2, analysis 7]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = 0.07, 90% CI 2-sided [-1.31 to 1.46], Standard Error of Mean 0.72
Statistical Analysis 11: Comparison: PF-06372865 17.5 mg vs Lorazepam 2 mg; [analysis description as in outcome 2, analysis 7]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -0.77, 90% CI 2-sided [-2.19 to 0.65], Standard Error of Mean 0.74
Statistical Analysis 12: Comparison: PF-06372865 52.5 mg vs Lorazepam 2 mg; [analysis description as in outcome 2, analysis 7]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -0.7, 90% CI 2-sided [-2.09 to 0.70], Standard Error of Mean 0.72
Statistical Analysis 13: Comparison: PF-06372865 17.5 mg vs Placebo; In eyes open condition. The same mixed model repeated measures analysis as applied to the primary outcome measure was used; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -4.42, 90% CI 2-sided [-5.60 to -3.25], Standard Error of Mean 0.68
Statistical Analysis 14: Comparison: PF-06372865 52.5 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -4.37, 90% CI 2-sided [-5.57 to -3.17], Standard Error of Mean 0.69
Statistical Analysis 15: Comparison: Lorazepam 2 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -4.38, 90% CI 2-sided [-5.57 to -3.19], Standard Error of Mean 0.69
Statistical Analysis 16: Comparison: PF-06372865 17.5 mg vs PF-06372865 52.5 mg; [analysis description as in outcome 2, analysis 13]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-1.08 to 1.19], Standard Error of Mean 0.66
Statistical Analysis 17: Comparison: PF-06372865 17.5 mg vs Lorazepam 2 mg; [analysis description as in outcome 2, analysis 13]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = -0.04, 90% CI 2-sided [-1.18 to 1.10], Standard Error of Mean 0.66
Statistical Analysis 18: Comparison: PF-06372865 52.5 mg vs Lorazepam 2 mg; [analysis description as in outcome 2, analysis 13]; Test type: Other; Mixed Model Repeated Measures Analysis; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-1.11 to 1.13], Standard Error of Mean 0.65

3. Secondary Outcome: The Percentage of Participants With Complete Suppression, Partial Response, and no Response to Intermittent Photic Stimulation (IPS)
Description: Complete suppression: SPR = 0 in all three eye conditions at the same time point. Partial response: A reduction in SPR of at least 3 units from baseline for at least 3 time points, and no time points with at least 3 units of increase, in the most sensitive eye condition; without meeting the complete suppression definition. No response: Did not meet complete suppression or partial response definitions.
Time Frame: Pre-dose, 1, 2, 4 and 6 hours post-dose
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | PF-06372865 17.5 mg | PF-06372865 52.5 mg | Lorazepam 2 mg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 7
Percentage of participants
  Complete suppression | 85.7 | 85.7 | 85.7 | 28.6
  Partial response | 0 | 0 | 0 | 0
  No response | 14.3 | 14.3 | 14.3 | 71.4

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-06372865
Time Frame: 1, 2, 4 and 6 hours post-dose
Population: All enrolled participants treated who had at least 1 measureable concentration in the respective study dose period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06372865 17.5 mg | PF-06372865 52.5 mg
Number analyzed (Participants) | 7 | 7
ng/mL | 81.30 (23) | 200.6 (45)

5. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-06372865
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose
Population: All enrolled participants treated who had at least 1 measureable concentration in the respective study dose period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06372865 17.5 mg | PF-06372865 52.5 mg
Number analyzed (Participants) | 7 | 7
ng*hr/mL | 331.3 (22) | 771.4 (56)

6. Secondary Outcome: Time for Cmax (Tmax) of PF-06372865
Time Frame: 1, 2, 4 and 6 hours post-dose
Population: All enrolled participants treated who had at least 1 measureable concentration in the respective study dose period.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06372865 17.5 mg | PF-06372865 52.5 mg
Number analyzed (Participants) | 7 | 7
hour | 2.12 (22) [1.02 to 3.03] | 3.02 (56) [1.98 to 5.95]

7. Secondary Outcome: Plasma Concentration of Lorazepam
Time Frame: 1, 2, 3, 4 and 6 hours post-dose
Population: All enrolled participants treated who had at least 1 measureable concentration in the respective study dose period.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lorazepam 2 mg
Number analyzed (Participants) | 7
ng/mL
  1 hours post dose: number analyzed (Participants) | 5
  1 hours post dose | 7.38 (5.92)
  2 hours post dose | 13.32 (6.67)
  3 hours post dose | 17.10 (4.32)
  4 hours post dose | 17.87 (2.97)
  6 hours post dose | 15.93 (1.92)

8. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities
Description: Safety laboratory tests included hematological, clinical chemistry (serum) and urinalysis safety tests.
Time Frame: 17 weeks
Population: The Safety Analysis Set included all participants who received at least 1 dose of investigational product in the respective study treatment period.
Measure: Number; unit: Participants
Arm/Group | PF-06372865 17.5 mg | PF-06372865 52.5 mg | Lorazepam 2 mg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 7
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Blood Pressure and Pulse Rate
Time Frame: 17 weeks
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | PF-06372865 17.5 mg | PF-06372865 52.5 mg | Lorazepam 2 mg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 7
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Findings
Time Frame: 17 weeks
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | PF-06372865 17.5 mg | PF-06372865 52.5 mg | Lorazepam 2 mg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 7
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: The all causalities treatment-emergent AEs by System Organ Class and Preferred Term in >5% of subjects. AEs included serious AEs and non-serious AEs.
Time Frame: 19 weeks
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | PF-06372865 17.5 mg | PF-06372865 52.5 mg | Lorazepam 2 mg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 7
Participants
  Treatment-emergent non serious AEs | 4 | 6 | 6 | 5
  Treatment-emergent serious AEs | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 19 weeks
Arm/Group | Placebo | PF-06372865 17.5 mg | PF-06372865 52.5 mg | Lorazepam 2 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/7 | 6/7 | 6/7 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | PF-06372865 17.5 mg (N=7) | PF-06372865 52.5 mg (N=7) | Lorazepam 2 mg (N=7)
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 3 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 3 | 3 | 4 | 3
Euphoric mood (Psychiatric disorders) | 0 | 0 | 1 | 1
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.